CLINICAL TRIAL: NCT04073160
Title: TRIO Bladder: A Phase Ib Study of Durvalumab (MEDI 4736) Plus Tremelimumab Followed by Concurrent Durvalumab Plus Bladder Radiation, Based on Molecular Subtypes in Muscle-Invasive Bladder Cancer
Brief Title: TRIO Bladder: A Study of Durvalumab Plus Tremelimumab Followed by Concurrent Durvalumab Plus Bladder Radiation in Muscle-Invasive Bladder Cancer
Acronym: TRIO Bladder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study will not be completed. No participants were enrolled.
Sponsor: Daniel George, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102352
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Bladder Cancer
Keywords: Muscle-invasive bladder cancer; Decipher bladder test; Durvalumab; Tremelimumab; Bladder radiation; Urothelial carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decipher Bladder test subtype non-basal (Experimental): Subjects with localized muscle invasive urothelial carcinoma of the bladder, whose tumor is Decipher Bladder test subtype non-basal
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Radiation: Bladder radiation; Drug: Intravesicular Therapy
- Decipher Bladder test subtype basal and cisplatin-ineligible (Experimental): Subjects with localized muscle invasive urothelial carcinoma of the bladder, whose tumor is Decipher Bladder test subtype basal and the subject is cisplatin-ineligible
  Interventions: Drug: Tremelimumab; Drug: Durvalumab; Radiation: Bladder radiation; Drug: Intravesicular Therapy

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab and durvalumab will be administered in combination during cycles 1 and 2. Tremelimumab will be administered intravenously at a dose of 75 mg on cycle 1 day 1 and cycle 2 day 1. Cycles are 4 weeks long.
Drug: Durvalumab — Tremelimumab and durvalumab will be administered in combination during cycles 1 and 2. Durvalumab will be administered intravenously at a dose of 1500 mg on cycle 1 day 1 and cycle 2 day 1. Cycles are 4 weeks long.
  Eligible subjects may go on to receive a combination of durvalumab and bladder radiation during cycles 3 and 4. Durvalumab will be administered intravenously at a dose of 1500 mg on cycle 3 day 1 and cycle 4 day 1.
  At the completion of radiation, eligible subjects may continue to receive durvalumab for a maximum of one year from the date of their initial dose. Durvalumab will be administered intravenously at a dose of 1500 mg on the first day of each cycle.
  Other Names: Imfinzi
Radiation: Bladder radiation — During the durvalumab cycles 3 and 4, eligible subjects will receive 6.5 weeks of radiation to the bladder. Radiation will be administered at a dose of 64 Gy in daily 2 Gy fractions.
Drug: Intravesicular Therapy — Subjects will receive intravesicular therapy, if clinically indicated during cycles 5 and beyond of durvalumab administration. Intravesicular therapy will consist of BCG, gemcitabine, mitomycin or a similar drug, depending on institutional standards and treating provider's discretion.

SUMMARY:
The purpose of this study is to describe the safety and tolerability of Durvalumab plus Tremelimumab followed by concurrent Durvalumab plus bladder radiation in patients with localized muscle invasive urothelial carcinoma of the bladder, who are either Decipher-Non-Basal OR Decipher-Basal and cisplatin-ineligible. Eligible subjects will receive 2 cycles of Durvalumab plus Tremelimumab followed by imaging and cystoscopy. Subjects whose cancer responds or is stable will receive a combination of 2 cycles of Durvalumab plus 6.5 weeks of radiation to the bladder followed by imaging and a TURBT. Subjects whose cancer continues to respond and meets certain criteria will continue to receive Durvalumab for up to 12 months from initial dose or until the cancer recoccurs or progresses, whichever occurs earlier. During this time, subjects may also receive intravesicular therapy if clinically indicated. Subjects will be followed for 5 years from initial dose.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Age ≥ 18 years
3. Histologically or cytologically confirmed urothelial carcinoma of the bladder. Non-urothelial histologies and upper tract disease are excluded.
4. Has clinical stage T2-T4b, N0-3, M0 urothelial carcinoma
5. DECIPHER-Non-basal (Group A) OR DECIPHER-Basal but cisplatin-ineligible (Group B)

   a. Cisplatin-ineligible based on ≥1 of the following:

   i. CrCl <60 ml/min

   ii. Grade 2 hearing loss or peripheral neuropathy

   iii. ECOG performance status of 2
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. Life expectancy of at least 12 weeks
8. Body weight >30kg
9. Adequate normal organ and marrow function as defined below:

   1. Hemoglobin ≥ 8.0 g/dL and asymptomatic
   2. Absolute neutrophil count (ANC ≥1.5 x 109/L)
   3. Platelet count ≥100 x 109/L
   4. Serum bilirubin ≤ 1.5 x Institutional Upper Limit of Normal (ULN) (Note: This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.)
   5. AST/SGOT and ALT/SGPT ≤ 2.5 x ULN
   6. Measured creatinine clearance (CL) >30 mL/min
10. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they meet the requirements below.

    1. Women < 45 years of age would be considered post-menopausal if they underwent surgical sterilization (bilateral oophorectomy or hysterectomy.
    2. Women 45 to <50 years of age would be considered post-menopausal if they have been amenorrheic for 18 months or more following cessation of exogenous hormonal treatments, if they have a documented follicle-stimulating hormone levels in the post-menopausal range (> 40 mlU/mL) or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    3. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, if they have a documented follicle-stimulating hormone levels in the post-menopausal range (> 40 mlU/mL) or underwent surgical sterilization (bilateral oophorecomy, bilateral salpingectomy or hysterectomy).
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Subjects must not have any of the following:

1. Prior systemic chemotherapy for bladder cancer
2. Any prior treatment with CTLA-4, including tremelimumab PD-1 or PD-L1 including durvalumab checkpoint inhibitors
3. Administration of an investigational therapeutic within 28 days prior to Cycle 1, Day 1
4. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug.
5. Prior pelvic radiation that precludes bladder radiation
6. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
7. Prior cystectomy
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Duke Principal Investigator.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Duke Principal Investigator.
9. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
10. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
11. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
12. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
13. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
15. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
16. History of allogenic stem cell transplant
17. History of active primary immunodeficiency
18. Active infection including, clinical evidence of active tuberculosis (cough >2 weeks' duration, fevers, night sweats, weight loss, and/or abnormal lung imaging), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Receipt of live attenuated vaccine within 30 days prior to Cycle 1 Day 1. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab or tremelimumab and up to 30 days after the last dose of durvalumab or tremelimumab.
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
21. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
22. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
23. Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 90 days after the last dose of study drug(s)
  To describe the safety and tolerability of durvalumab plus tremelimumab followed by concurrent durvalumab plus bladder radiation in patients as assessed by CTCAE version 5.0.
Incidence of serious adverse events | Up to 90 days after the last dose of study drug(s)
  To describe the safety and tolerability of durvalumab plus tremelimumab followed by concurrent durvalumab plus bladder radiation in patients as assessed by CTCAE version 5.0.
Incidence of adverse events of special interest | Up to 90 days after the last dose of study drug(s)
  To describe the safety and tolerability of durvalumab plus tremelimumab followed by concurrent durvalumab plus bladder radiation in patients as assessed by CTCAE version 5.0.
Incidence of adverse events leading to study drug discontinuation | Up to 90 days after the last dose of study drug(s)
  To describe the safety and tolerability of durvalumab plus tremelimumab followed by concurrent durvalumab plus bladder radiation in patients as assessed by CTCAE version 5.0.
Incidence of deaths | Up to 90 days after the last dose of study drug(s)
  To describe the safety and tolerability of durvalumab plus tremelimumab followed by concurrent durvalumab plus bladder radiation in patients as assessed by CTCAE version 5.0.

SECONDARY OUTCOMES:
2-year disease-free survival (DFS) for Decipher test sub-type basal vs. Decipher test sub-type non-basal | 2 years
  2-year disease-free survival (DFS) for Decipher test sub-type basal vs. Decipher test sub-type non-basal
Pathologic complete response rate on post-duravalumab/radiation TURBT | Cycle 4 Day 21
  Proportion of subjects with a pathologic complete response rate on post-duravalumab/radiation TURBT
Rate of salvage cystectomy | 5 years
  Proportion of subjects undergoing a salvage cystectomy after discontinuing study drug(s)
5-year disease-free survival (DFS) | 5 years
  Proportion of subjects remaining disease-free at 5 years
5-year overall survival (OS) | 5 years
  Proportion of subjects alive at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tian Zhang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No